CLINICAL TRIAL: NCT05556824
Title: A Multi-Center Study of Panosyl-Isomaltooligosaccharides (PIMO) Adjunctive to Proton Pump Inhibitor (PPI) Therapy to Treat Gastroesophageal Reflux Disease (GERD) in Subjects Who Are PPI-Responders or PPI-Partial Responders
Brief Title: Multi-Center Study of Panosyl-Isomaltooligosaccharides Adjunctive to PPI Therapy to Treat GERD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Microbiome Health Sciences (Industry)
Collaborators: VBHRC Virginia Catalyst (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHS-1031-04
Record Dates: First submitted 2022-09-21; First posted 2022-09-27 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gastroesophageal Reflux
Keywords: GERD; microbiome; PIMO; PPI; Heartburn; Gastroesophageal Reflux; Prebiotic
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug Product (Active Comparator): Panosyl-isomaltooligosaccharide (PIMO) liquid 1 g (1.5 ml) per day for 8 weeks
  Interventions: Drug: MHS-1031
- Placebo (Placebo Comparator): Placebo liquid (1.5 ml) per day for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MHS-1031 — Study medication will be supplied as a syrup in individual sachets containing 1g (1.5 mL) of MHS-1031. Subjects will be randomized in 2:1 fashion to either study drug (2) or placebo (1)
  Other Names: Panosyl-isomaltooligosaccharide
  Arms: Drug Product
Other: Placebo — Matching placebo is an oral solution formulated to have a degree of sweetness and acidity similar to the study medication and will be provided in equivalent sachets containing 1.5g (1.5 mL) of the oral placebo solution.
  Arms: Placebo

SUMMARY:
This study will be conducted as a multi-center, randomized, double-blind, placebo-controlled trial to evaluate the effect of MHS-1031 on heartburn-free days in subjects with GERD-related heartburn symptoms.

DETAILED DESCRIPTION:
MHS-1031 is a specific proprietary digestion-resistant oligosaccharide carbohydrate that serves as a prebiotic.

This study will be conducted as a multi-center, randomized, double-blind, placebo-controlled trial to evaluate the effect of MHS-1031 adjunctive to PPI therapy on heartburn-free days in subjects with GERD-related heartburn symptoms who self-report improvement while on sustained daily PPI therapy. Heartburn-free days will be determined by subject report specific to any of the three questions ("burning feeling behind the breastbone" and/or "pain behind your breastbone" and/or "heartburn"; Questions 1, 2 & 3 of the RESQ-eD). For purposes of this trial, heartburn-free days are defined as subject report of 'Did Not Have', or 'Very Mild' on each of the three RESQ-eD questions listed above.

All candidate subjects must self-report at least partial response to sustained daily PPI acid suppressive therapy (i.e. 'daily' defined as taking PPIs 5-7 days/week on average). Candidate subjects will be screened for medical history of chronic heartburn that may be associated with other medical conditions, and these subjects will be excluded. The entire study consists of three phases: Remote Screening Phase 2-Week Assessment (SP1), on-site Screening Phase Part 2 (SP2) and Treatment Phase (TP).

Efficacy will be assessed using patient reported outcome (PRO) questionnaires, concomitant medication assessments, and assessment of adverse events, from baseline (determined during Remote Screening Phase 2-Week Assessment) to Treatment Phase Weeks 1-4 and Weeks 5-8. The primary analyses will be conducted to assess the efficacy of MHS-1031 adjunctive to PPI therapy, and separately as monotherapy subsequent to combined PPI and MHS-1031 therapy, in randomized subjects with GERD-related heartburn as determined by the RESQ-eD validated questionnaire, validated for use online.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator or sub-investigators, the subject is capable of understanding and complying with protocol requirements, including compliance with completing nightly online questionnaires in one of the IRB-approved languages.
* Subject signs and dates an electronic (Screening Phase Part 1) and site-specific written informed consent form (ICF) and any required privacy authorization prior to the initiation of any study procedures.
* Ability, during Remote Screening Phase 2-Week Assessment, to complete all required online nightly RESQ-eD questionnaires, medication questionnaires, 4-item Patient Health Questionnaire for Depression and Anxiety (PHQ-4) questionnaire and Participant Global Assessment questionnaire.
* Access to a computer/tablet/phone with internet access and active email account in order to complete online questionnaires daily throughout study participation.
* Males or females ≥18 and ≤75 years of age, with a BMI ≥ 18 and < 35 kg/m2.
* Female subjects must be postmenopausal or surgically sterile or, if of childbearing potential, must agree to use a medically acceptable form of contraception from the time of signing the informed consent form through completion of study. If only the barrier method is used, a single barrier or better is adequate. Postmenopausal women must have had ≥ 12 months of spontaneous amenorrhea. Surgically sterile women are defined as those who have had a hysterectomy, bilateral ovariectomy, or bilateral tubal ligation. All women of childbearing potential must have a negative pregnancy test result before administration of study drug.
* Must be on stable doses of medications, if any, prescribed for chronic conditions other than GERD.
* Subject must be taking daily PPI (defined as 5-7 days/week on average) for at least four (4) consecutive weeks with self-reported symptom improvement (frequency and/or severity) prior to the Screening Call selected from the following list of medications:
* omeprazole
* esomeprazole
* lansoprazole
* dexlansoprazole
* pantoprazole
* rabeprazole
* Onset of GERD-related heartburn symptoms for a minimum of 3 months prior to Screening Call (i.e., "burning feeling behind the breastbone" and/or "pain behind your breastbone" and/or "heartburn" per questions 1, 2 or 3 of RESQ-eD).
* Subject has maintained a stable diet and exercise regimen for ≥ 30 days prior to the Screening Call and is willing to maintain that diet and exercise regimen for the duration of the study (i.e., if subject is currently following diets including, but not limited to, Keto, FODMAP, Vegan, Vegetarian, s/he must be willing to continue this dietary lifestyle through end-of-study visit).

Exclusion Criteria:

* Current use of any mouthwash (e.g., Listerine, Scope, others) or unwilling to discontinue use for the duration of the study (requires 3-day washout prior to starting the Remote Screening Phase 2-Week Assessment)
* Teeth whitening within 7 days of Screening Call or current use of teeth whitening substances (not including teeth whitening toothpaste) or unwilling to discontinue use for the duration of the study (requires 7-day washout prior to starting the Remote Screening Phase 2-Week Assessment).
* Current use of histamine 2 receptor antagonists (H2RAs) (requires 7-day washout prior to starting the Remote Screening Phase 2-Week Assessment).
* Surgical procedure requiring general anesthesia within 60 days of the Screening Call
* Colonoscopy, high colonic, colonic cleanse or barium enema in the past 30 days, or scheduled for colonoscopy or barium enema at any time for the duration of the study, and unwilling to postpone until after study completion.
* History of cancer diagnosis and/or treatment (other than basal cell carcinoma of the skin) within the preceding five (5) years.
* Concomitant illness with potential to confound outcome assessments for this study, including, but not limited to:

  * History of untreated peptic or gastric ulcer, Zollinger-Ellison syndrome, or Helicobacter pylori (H. pylori) positivity without a history of successful treatment
  * History of ulcerative colitis or Crohn's disease.
  * Stomach ulcers, pancreaticobiliary disorder (e.g., gallstones bile duct stones, pancreatic stones, pancreatitis), diverticulitis symptomatic within the past 6 months.
* Acute or chronic hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection.
* Significant current morbidity of the heart, kidney, liver or lung.
* History of Long QT Syndrome
* History of Torsades de pointes (TdP)
* Current neurological or psychiatric disorder (e.g., Parkinson's, Huntington's chorea, schizophrenia, seizure, bi-polar disorder, major depressive disorder).
* Known or suspected alcoholism, drug addiction, or significant drug abuse within 1 year of the Screening Call based on subject reporting and PI assessment.
* Active history of tobacco or nicotine use (of any type) in the last 6 months averaging more than 1 cigar/cigarette per week. Vaping products and e-cigarettes that contain nicotine and/or tobacco are not allowed. Chewing tobacco and nicotine gum are prohibited at any level. Nicotine patches are NOT exclusionary.
* Alcohol abuse (for alcohol defined as: > 14 drinks/week or 4 drinks/day for men, 7 drinks/week or 3 drinks/day for women).
* Intake of acetylsalicylic acid (i.e., aspirin) at doses > 162 mg/day.
* Non-steroidal anti-inflammatory pain relievers (NSAIDs) such as ibuprofen (Advil®, Motrin® IB, others) >/= 4 days/week on average not to exceed half the recommended maximum prescription daily dosing as listed in the Physician's Desk Reference.
* Acetaminophen > 2,000 mg/day
* Inhalation or ingestion of products containing delta-9-tetrahydrocannabinol (THC) > 2 days/week on average.
* Any known medical condition, clinical signs and symptoms, vital signs, abnormal laboratory, or other testing that are not well controlled on stable dosing of medication for at least 90 days prior to the Screening Call or are considered clinically significant by the Principal Investigator (PI), that could interfere with the subject's participation in and completion of the study. Examples of medical conditions including, but not limited to:
* Uncontrolled hypertension
* Uncontrolled diabetes
* History of adrenal disease, diabetic nephropathy, or gastroparesis
* Uncontrolled hypothyroidism
* Untreated mental disorder
* Paraplegia or Quadriplegia
* Cerebrovascular event (stroke) or myocardial infarction (MI) within the last 6 months.
* Structural abnormality of the GI tract, or disease or condition that can affect GI motility (e.g., achalasia, esophageal atresia), or defecation.
* Planned travel outside the US during the study period or routine travel within the US during the study period that results in >2-hour time zone difference.
* Cyclical work shift (e.g., routinely switching between day shifts and night shifts)
* Any of the following current (within the past 6 months) symptomatic conditions:

  * pseudo-obstruction,
  * malignant polyps (requiring surgery),
  * abdominal adhesions confirmed via laparoscopy,
  * intestinal ischemia without colitis,
  * laxative or enema abuse.
* History of ischemic colitis in the past 5 years.
* Current COVID19 infection, or a history of a prior COVID19 infection with ongoing symptoms suggestive of "Long COVID".
* Endoscopic evidence of any of the following:

  * Eosinophilic esophagitis, scleroderma, Barrett's esophagus, esophageal cancer, Candida esophagitis confirmed by histopathology.
  * LA grade B, C, or D erosive esophagitis, esophageal stricture or scarring.
  * History of surgery or endoscopic treatment including fundoplication and/or dilation for esophageal stricture.
* History of fecal impaction that required hospitalization or emergency room treatment within 3 months of the Screening Call.
* History of eating disorder within the last 2 years.
* Symptomatic condition (e.g., polycystic kidney disease, endometriosis, ovarian cysts, etc.) during the 12 months prior to the Screening Call that required intervention (i.e., clinic or emergency room visit or hospitalization) that may be associated with chronic abdominal pain or discomfort and might confound the assessments in this study.
* Surgical history that meets any of the following criteria:
* Gastric bypass surgery or invasive procedure for the treatment of obesity or surgery to remove a segment of the GI tract at any time prior to the Screening Call
* Gastric band present within the past 60 days
* Open surgery of the abdomen, pelvis, or retroperitoneal structures within 6 months prior to the Screening Call
* Laparoscopic appendectomy or cholecystectomy or other instrumentation of the bowel < 60 days prior to the Screening Call. NOTE: Endoscopic removal of benign polyps is not exclusionary.
* Prior use of the study medication MHS-1031 or ISOThrive Prebiotic Nectar.
* Use of fructo-oligosaccharides (FOS) or inulin.
* Symptomatic condition (e.g., angina, rumination, or other conditions involving the mouth and/or throat) during the 12 months prior to the Screening Call.
* Use of any of the following medications that have not been stable dosing for at least 90 days at time of Screening Call:

  * Anticholinergics, such as oxybutynin (e.g., Ditropan XL®)
  * Theophylline (e.g., Elixophyllin®, Theochron)
  * Bisphosphonates taken orally, such as alendronate (Fosamax), ibandronate (Boniva) and risedronate (Actonel®, Atelvia®)
  * Quinidine
  * Anticoagulants (e.g., Coumadin, Heparin)
  * Iron supplement (other than contained in multi-vitamin)
  * Potassium supplements in pill form (Elixirs are NOT exclusionary)
  * Asthma medications
  * Prescription medication to control Irritable Bowel Syndrome or Chronic Idiopathic Constipation
* Use of Nitrates within the last 12 months.
* Medication for depression, anxiety, or sleep (e.g., benzodiazepines such as diazepam (Valium®) and temazepam (Restoril) with uncontrolled symptoms or medication dosing that has not been stable for at least 90 days at time of Screening Call.
* Antibiotic use within 60 days of the Screening Call.
* Narcotic (e.g., opiate) or illicit drug (i.e., illegal at both the Federal and State levels; e.g. Cocaine, Heroin, Methamphetamine) use within 60 days of the Screening Call.
* Use of any investigational product within 90 days prior to the Screening Call.
* Use of GLP-1 agonists (e.g., Dulaglutide (Trulicity), Exenatide, Semaglutide (Ozempic/Wegovy), Liraglutide) or prescription medications used for weight loss within 6 months of Screening Call.

  * Current use of potassium-competitive acid blocker (PCAB). PCAB may not be used within one week of screening call.
* Pregnancy, lactation, planned pregnancy or planned ova donation during the study period.
* Participation in another investigation (clinical trial) during the course of this study.
* Any major lifestyle change, such as getting married, change in residence, change in job, or other highly stressful event planned during the study periods.
* Sustained daily use of PPIs without self-report of improvement of heartburn symptoms.
* Self or relative employed directly or indirectly by the Sponsor or relative or employee of investigator or investigator's staff.
* Other conditions or situations that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Heartburn-free days/week | 4 and 8 weeks
  The difference between baseline weekly average heartburn-free days and weekly average heartburn-free days during Treatment Phase Weeks 1-4 and Weeks 5-8 (as measured using questions 1, 2 and 3 of the Reflux Symptom Questionnaire Electronic Diary) (RESQ-eD).

SECONDARY OUTCOMES:
Heartburn symptom severity | 4 and 8 weeks
  The difference between baseline daily average heartburn symptom severity score and daily average heartburn symptom severity score during Treatment Phase Weeks 1-4 and Treatment Phase Weeks 5-8 (as measured using questions 1, 2 and 3 of the Reflux Symptom Questionnaire Electronic Diary) (RESQ-eD).
Heartburn-free day satisfaction | 4 and 8 weeks
  Any increase between baseline weekly average heartburn-free days and heartburn-free days during Treatment Phase Weeks 1-4 and Weeks 5-8 where Patient Global Assessment Question 1 is ≥ baseline.
GERD-related severity satisfaction | 4 and 8 weeks
  Any increase between baseline daily average heartburn severity and heartburn severity during Treatment Phase Weeks 1-4 and Weeks 5-8 where Patient Global Assessment Question 1 is ≥ baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Swann, MD, Principal Investigator — Microbiome Health Sciences
Locations (18):
- United States (18):
  - Elite Clinical Studies LLC, Phoenix, Arizona
  - Angel City Research, Los Angeles, California
  - Wr-Msra, Llc, Lake City, Florida
  - A Positive Clinical Research, Miami, Florida
  - Advanced Gastroenterology Associates LLC, Palm Harbor, Florida
  - Health Synergy Clinical Research, West Palm Beach, Florida
  - West Palm Quality Research (WPQR), West Palm Beach, Florida
  - EmVenio-Georgia (EMGA), Atlanta, Georgia
  - WR-Mount Vernon Clinical Research (MVCR), Sandy Springs, Georgia
  - Gastroenterology Associates of Western Michigan PLC (WMCR), Wyoming, Michigan
  - M3 Wake Research (CPOR), Raleigh, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - SMS Clinical Research (SMSR), Mesquite, Texas
  - A and U Family Medicine (NCR), Sugar Land, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Charlottesville Medical Research Center, Charlottesville, Virginia
  - Digestive Disease and Liver Specialists, Norfolk, Virginia
  - GI Research Partners, LLC, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No